CLINICAL TRIAL: NCT00074412
Title: A Phase III Trial to Determine the Efficacy and Safety of an Extended Regimen of Nevirapine in Infants Born to HIV-Infected Women to Prevent Vertical HIV Transmission During Breastfeeding
Brief Title: Using Nevirapine to Prevent Mother-to-Child HIV Transmission During Breastfeeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HPTN 046; 10142 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2003-12-11; First posted 2003-12-15 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 2A (Experimental): For infants: extended treatment with NVP
  Interventions: Drug: Nevirapine
- 2B (Placebo Comparator): For infants: extended treatment with NVP placebo
  Interventions: Drug: Nevirapine placebo

INTERVENTIONS:
Drug: Nevirapine — 10 mg/ml oral suspension taken once daily up to 6 months of age. Dosage will increase throughout study.
  Other Names: NVP
  Arms: 2A
Drug: Nevirapine placebo — Oral suspension taken once daily up to 6 months of age
  Other Names: NVP placebo
  Arms: 2B

SUMMARY:
The many benefits of breastfeeding are well documented. However, because of the risk of mother-to-child transmission (MTCT) of HIV from an HIV infected mother to her infant, there is considerable concern over the practice, especially in developing countries. The purpose of this study is to determine the safety and effectiveness of the anti-HIV drug nevirapine (NVP) in preventing MTCT of HIV in breastfeeding infants born to HIV infected women in South Africa, Tanzania, Uganda, and Zimbabwe.

DETAILED DESCRIPTION:
Breastfeeding provides general health, growth, and development benefits to an infant and significantly decreases the risk of certain acute and chronic diseases. Breastfeeding also decreases financial burden on the mother by decreasing the need for infant formula and health care for the infant. However, clinical evidence has shown that HIV can be readily transmitted through breast milk, although the risk of HIV MTCT over time while breastfeeding has been difficult to determine. Given the many advantages of breastfeeding and the significant obstacles to substituting formula for breast milk in developing countries, there is an urgent need to make breastfeeding by HIV infected women safe. This study will evaluate the safety and efficacy of an extended NVP regimen for prevention of MTCT of HIV through breastfeeding.

This study will last approximately 3.5 years. Mother/infant pairs will be enrolled over a period of 18 to 24 months. During the third trimester of pregnancy, HIV infected participants will receive HIV counseling and the intrapartum/neonatal two-dose NVP prophylaxis regimen to prevent MTCT. Mothers will also be given infant feeding options counseling and information on administering the study drug to the infant. Infants who were randomly assigned to receive a placebo and older than 6 weeks of age as of 08/10/07 OR to receive NVP will continue their treatment assignment. Infants who were randomly assigned to receive a placebo and are 6 weeks of age or less as of 08/10/07 will receive open-label NVP through Day 42 of life. For all other participants, all randomized infants will receive extended NVP through 6 weeks (Day 42) of life. All eligible infants will be randomly assigned to one of two groups at Week 6 following birth. The first group will receive extended NVP treatment; the second group will receive nevirapine placebo. Randomized infants will receive the extended NVP or NVP placebo through the first 6 months of life or until cessation of breastfeeding, whichever occurs earlier. Mothers will be instructed to begin giving their infants their assigned intervention starting at Day 3 to Day 7 postpartum. All mothers and infants outside of the study will be offered the local standard of care antiretroviral (ARV) regimen for the prevention of MTCT, but these ARVs will not be provided by the study.

Follow-up evaluations will be conducted at Weeks 2 and 6 and Months 3, 6, 12, and 18 for mothers, and at Weeks 2, 5, 6, and 8 and Months 3, 4, 5, 6, 9, 12, and 18 for infants. Study visits will include physical examinations, blood tests (including HIV tests), and medical histories. Study participants will be followed for up to 3.5 years.

ELIGIBILITY:
Note: As of 08/10/07, the arm assignments for current and new participants have changed. Please see the above description for this trial for more information.

Inclusion Criteria for Mothers:

* 18 years of age or older
* HIV infected
* In third trimester of pregnancy, or at most 3 days post-delivery
* If baby is not yet born, planning to deliver at a facility where the study is being conducted
* Plan to breastfeed

Exclusion Criteria for Mothers:

* Complications with this pregnancy
* Serious medical condition that would interfere with the study (e.g., that would prevent breastfeeding or adherence to the follow-up schedule), as judged by the on-site clinician

Inclusion Criteria for Infants:

* Born to an HIV infected mother who is eligible for the study
* Weighed at least 2000 grams (4.4 lbs) at birth
* Blood sample obtained from the infant for HIV-1 DNA PCR, CBC with differential, and ALT
* Infants in a multiple birth are eligible only if both/all infants are eligible for the study and assigned to the same study group
* Able to breastfeed (e.g., mother and infant alive with no condition apparent that would prevent breastfeeding)

Exclusion Criteria for Infants:

* HIV DNA PCR positive at birth
* ALT of Grade 2 or higher at birth
* Hemoglobin, absolute neutrophil count, or platelet count of Grade 3 or higher at birth
* Skin rash of Grade 2B (urticaria), Grade 3, or above
* Confirmed or suspected clinical hepatitis
* Serious illness or condition that would interfere with compliance with study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2026 (Actual)
Dates: Start 2007-01; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoosen M. Coovadia, MD, MBBS, Study Chair — Centre for HIV Networking (HIVAN), Nelson Mandela School of Medicine, University of Natal; Laura Guay, MD, Study Chair — Johns Hopkins University; Wafaie Fawzi, MD, PhD, Study Chair — Department of Nutrition, Harvard School of Public Health; Yvonne Maldonado, MD, Study Chair — Stanford University; Daya Moodley, MSc, PhD, Study Chair — Department of Obstetrics and Gynaecology, Nelson R Mandela School of Medicine, University of Natal
Locations (5):
- CAPRISA Umlazi CRS, Umlazi, KwaZulu-Natal, South Africa
- Muhimbili University of Health and Allied Sciences (MUHAS) CRS, Dar es Salaam, Tanzania
- Makerere University- JHU Research Collaboration {MUJHU CARE LTD} CRS, Kampala, Mpigi, Uganda
- Zimbabwe (2):
  - Seke North CRS, Chitungwiza
  - St Mary's CRS, Chitungwiza

REFERENCES:
- [Background] Jackson JB, Musoke P, Fleming T, Guay LA, Bagenda D, Allen M, Nakabiito C, Sherman J, Bakaki P, Owor M, Ducar C, Deseyve M, Mwatha A, Emel L, Duefield C, Mirochnick M, Fowler MG, Mofenson L, Miotti P, Gigliotti M, Bray D, Mmiro F. Intrapartum and neonatal single-dose nevirapine compared with zidovudine for prevention of mother-to-child transmission of HIV-1 in Kampala, Uganda: 18-month follow-up of the HIVNET 012 randomised trial. Lancet. 2003 Sep 13;362(9387):859-68. doi: 10.1016/S0140-6736(03)14341-3. PMID 13678973
- [Background] Mitchla Z, Sharland M. Current treatment options to prevent perinatal transmission of HIV. Expert Opin Pharmacother. 2000 Jan;1(2):239-48. doi: 10.1517/14656566.1.2.239. PMID 11249545
- [Background] Mofenson LM. Advances in the prevention of vertical transmission of human immunodeficiency virus. Semin Pediatr Infect Dis. 2003 Oct;14(4):295-308. doi: 10.1053/j.spid.2003.09.003. PMID 14724794
- [Background] Piwoz EG, Ross J, Humphrey J. Human immunodeficiency virus transmission during breastfeeding: knowledge, gaps, and challenges for the future. Adv Exp Med Biol. 2004;554:195-210. PMID 15384577
- [Derived] Bhattacharya D, Guo R, Tseng CH, Emel L, Sun R, Zhang TH, Chiu SH, Stranix-Chibanda L, Chipato T, Ship H, Mohtashemi NZ, Kintu K, Manji KP, Moodley D, Maldonado Y, Currier JS, Thio CL. Hepatitis B virus clinical and virologic characteristics in an HIV perinatal transmission study in sub-Saharan Africa. AIDS. 2024 Mar 1;38(3):329-337. doi: 10.1097/QAD.0000000000003752. Epub 2023 Oct 17. PMID 37861675
- [Derived] Bhattacharya D, Guo R, Tseng CH, Emel L, Sun R, Chiu SH, Stranix-Chibanda L, Chipato T, Mohtashemi NZ, Kintu K, Manji KP, Moodley D, Thio CL, Maldonado Y, Currier JS. Maternal HBV Viremia and Association With Adverse Infant Outcomes in Women Living With HIV and HBV. Pediatr Infect Dis J. 2021 Feb 1;40(2):e56-e61. doi: 10.1097/INF.0000000000002980. PMID 33181788
- [Derived] Nandlal V, Moodley D, Grobler A, Bagratee J, Maharaj NR, Richardson P. Anaemia in pregnancy is associated with advanced HIV disease. PLoS One. 2014 Sep 15;9(9):e106103. doi: 10.1371/journal.pone.0106103. eCollection 2014. PMID 25222119
- [Derived] Fowler MG, Coovadia H, Herron CM, Maldonado Y, Chipato T, Moodley D, Musoke P, Aizire J, Manji K, Stranix-Chibanda L, Fawzi W, Chetty V, Msweli L, Kisenge R, Brown E, Mwatha A, Eshleman SH, Richardson P, Allen M, George K, Andrew P, Zwerski S, Mofenson LM, Jackson JB; HPTN 046 Protocol Team. Efficacy and safety of an extended nevirapine regimen in infants of breastfeeding mothers with HIV-1 infection for prevention of HIV-1 transmission (HPTN 046): 18-month results of a randomized, double-blind, placebo-controlled trial. J Acquir Immune Defic Syndr. 2014 Mar 1;65(3):366-74. doi: 10.1097/QAI.0000000000000052. PMID 24189151
- [Derived] Coovadia HM, Brown ER, Fowler MG, Chipato T, Moodley D, Manji K, Musoke P, Stranix-Chibanda L, Chetty V, Fawzi W, Nakabiito C, Msweli L, Kisenge R, Guay L, Mwatha A, Lynn DJ, Eshleman SH, Richardson P, George K, Andrew P, Mofenson LM, Zwerski S, Maldonado Y; HPTN 046 protocol team. Efficacy and safety of an extended nevirapine regimen in infant children of breastfeeding mothers with HIV-1 infection for prevention of postnatal HIV-1 transmission (HPTN 046): a randomised, double-blind, placebo-controlled trial. Lancet. 2012 Jan 21;379(9812):221-8. doi: 10.1016/S0140-6736(11)61653-X. Epub 2011 Dec 22. PMID 22196945
- [Derived] Aizire J, Fowler MG, Wang J, Shetty AK, Stranix-Chibanda L, Kamateeka M, Brown ER, Bolton SG, Musoke PM, Coovadia H. Extended prophylaxis with nevirapine and cotrimoxazole among HIV-exposed uninfected infants is well tolerated. AIDS. 2012 Jan 28;26(3):325-33. doi: 10.1097/QAD.0b013e32834e892c. PMID 22112598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-infected pregnant women were recruited from antenatal clinics at DAIDS Clinical Trials Sites in Zimbabwe, South Africa, Uganda & Tanzania between May 14, 2008 & January 20th 2010. 1700 mother/infant pairs were enrolled & infants were given daily doses of Nevirapine for 6 weeks at which point there were randomized to placebo or extended NVP.
Pre-assignment Details: Infants were excluded from randomization if in first 42 days: had a positive HIV-1 DNA PCR, breastfeeding was discontinued, never initiated or permanently discontinued open-label NVP, certain graded abnormal labs, skin rash grade2B or higher, clinical hepatitis, serious illness/condition that prevented compliance, or use of rifampin/ketoconazole.
Groups:
- Placebo: For infants: extended treatment with NVP placebo
- Nevirapine: For infants: extended treatment with NVP
Period: Overall Study
Arm/Group | Placebo | Nevirapine
Started | 763 (Number of infants randomized at 6 weeks.) | 759 (Number of infants randomized at 6 weeks.)
Week 8 Visit | 759 | 759
Month 3 Visit | 759 | 755
Month 4 Visit | 758 | 752
Month 5 Visit | 756 | 750
Month 6 Visit | 748 | 748
Month 9 Visit | 741 | 741
Month 12 Visit | 733 | 735
Completed | 681 (Number of infants who completed final 18 month visit: out of 733 infants who were expected.) | 675 (Number of infants who completed final 18 month visit: out of 733 infants who were expected.)
Not Completed | 82 | 84
Not completed — Death | 30 | 26
Not completed — Lost to Follow-up | 52 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nevirapine | Placebo | Total
Number analyzed (Participants) | 759 | 763 | 1522
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 759 | 763 | 1522
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Ambiguous | 1 | 0 | 1
  Male | 363 | 398 | 761
  Female | 395 | 365 | 760
Region of Enrollment [Number; unit: participants]
  Tanzania | 98 | 99 | 197
  Uganda | 259 | 261 | 520
  South Africa | 171 | 171 | 342
  Zimbabwe | 231 | 232 | 463
Categorical Infant Birthweight (g) [Number; unit: participants]
  Missing | 0 | 1 | 1
  2000-2499 | 50 | 52 | 102
  2500-2999 | 214 | 211 | 425
  3000-3499 | 329 | 336 | 665
  >=3500 | 166 | 163 | 329

OUTCOME MEASURES:

1. Primary Outcome: HIV Infection in Infants Determined to be HIV Uninfected at 6 Weeks Enrolled in Each Arm of the Study
Time Frame: At Month 6
Population: All infants who were randomly allocated to either treatment or placebo at 6 weeks of age under version 3.0 of the protocol were included in the analysis of the primary endpoint, HIV infection at 6 months. 127/1700 infants were enrolled but excluded from randomization at 6 weeks for various reasons as mentioned in the flow-through.
Measure: Number; unit: participants
Arm/Group | Nevirapine | Placebo
Number analyzed (Participants) | 759 | 763
participants
  # of HIV infections at 6 months | 8 [0.3 to 1.9] | 18 [1.3 to 3.6]
  # of Infants at risk for HIV infection at 6 months | 700 | 699
Statistical Analysis 1: Comparison: Nevirapine; Test type: Superiority or Other; Kaplan-Meier Method; 6 month Rate of Cum. HIV Infection (%) = 1.1, 95% CI 2-sided [0.3 to 1.8]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; Kaplan-Meier Method; 6 month Rate of Cum. HIV Infection (%) = 2.4, 95% CI 2-sided [1.3 to 3.6]
Statistical Analysis 3: Comparison: Nevirapine vs Placebo; Assuming the cumulative HIV infection rate in placebo group would be 4.2% (2.6 at 6 wk. & 6.7 at 6 mon.), we estimated 1500 mother/infant pairs would provide 90% power to detect a reduction in HIV infection from 4.2% to 1.4% at 6 mon. with a Pearson χ² test statistic and a one-sided false positive error rate of 0.025. Rate of cumulative infection was calculated using Kaplan-Meier method and rates between extended NVP group and placebo were done with the Z statistic; Test type: Superiority or Other; p = 0.049, Z-test — P-value has not been adjusted for interim analysis or multiple testing. A priori threshold for statistical significance was 0.05; Z statistic = 1.973

2. Primary Outcome: Frequency and Severity of Adverse Reactions Among Participating Infants
Description: For those infants who were randomized at 6 weeks and who initiated study drug we looked at the frequency and severity of adverse reactions through 18 months of study. The severity of all AEs was graded according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. The term severity is described as the intensity grade or level for specific event (i.e. mild, moderate, severe, or life-threatening). Severity is not the same as seriousness.
Time Frame: 6 weeks through 18 months
Population: A total of 1519 infants, 758 in the NVP arm and 761 in the placebo arm, initiated study product and were thus included in the analysis for the frequency and severity of adverse reactions.
Measure: Number; unit: Number of Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Nevirapine | Placebo
Number analyzed (Participants) | 758 | 761
Number analyzed (Adverse Events) | 2014 | 1964
Number of Adverse Events
  Death | 26 | 30
  Life-Threatening | 87 | 87
  Severe | 375 | 332
  Moderate | 694 | 677
  Mild | 832 | 838

3. Secondary Outcome: Proportion of Infants Who Are Alive and HIV-uninfected in the Two Arms
Time Frame: At Months 6 and 18
Population: There were 1522 infants randomized at 6 weeks of birth to either the extended Nevirapine arm (759) or the placebo arm (763).
Measure: Number; unit: participants
Arm/Group | Nevirapine | Placebo
Number analyzed (Participants) | 759 | 763
participants
  Number of Infants Alive and HIV-free at 6 months | 689 | 683
  Number of Infants Alive and HIV-free at 18 months | 629 | 616
Statistical Analysis 1: Comparison: Nevirapine; The cumulative rate of HIV-free survival at 6 months in the extended NVP arm was calculated using the Kaplan-Meier method; while the 95% CI was calculated using Greenwood's formula; Test type: Superiority or Other; Kaplan-Meier Method; Cum. Rate of HIV-free Survival 6mon (%) = 97.7, 95% CI 2-sided [96.6 to 98.8]
Statistical Analysis 2: Comparison: Placebo; The cumulative rate of HIV-free survival at 6 months in the placebo arm was calculated using the Kaplan-Meier method; while the 95% CI was calculated using Greenwood's formula; Test type: Superiority or Other; Kaplan-Meier Method; Cum. Rate of HIV-free Survival 6mon (%) = 96.8, 95% CI 2-sided [95.5 to 98.0]
Statistical Analysis 3: Comparison: Nevirapine vs Placebo; The cumulative rates of HIV-free survival at 6 months were compared between the two groups using a Z-statistic; Test type: Superiority or Other; p = 0.274, Z-test — P-value was not adjusted for interim analysis or multiple testing; Z statistic = 1.095
Statistical Analysis 4: Comparison: Nevirapine; The cumulative rate of HIV-free survival at 18 months in the extended NVP arm was calculated using the Kaplan-Meier method; while 95% confidence intervals were calculated using Greenwood's formula; Test type: Superiority or Other; Kaplan-Meier Method; Cum. Rate of HIV-free Survival 18mon (%) = 94.5, 95% CI 2-sided [92.9 to 96.2]
Statistical Analysis 5: Comparison: Placebo; The cumulative rate of HIV-free survival at 18 months in the placebo arm was calculated using the Kaplan-Meier method; while the 95% confidence interval was calculated using Greenwood's formula; Test type: Superiority or Other; Kaplan-Meier Method; Cum. Rate of HIV-free Survival 18mon (%) = 93.3, 95% CI 2-sided [91.5 to 95.1]
Statistical Analysis 6: Comparison: Nevirapine vs Placebo; The cumulative rates of HIV-free survival at 18 months were compared between the two groups using a Z statistic; Test type: Superiority or Other; p = 0.323, Z-test — P-value was not adjusted for interim analysis or multiple testing; Z statistic = 0.988

4. Secondary Outcome: Relative Rates of HIV Infection in the Two Arms
Time Frame: At Month 18
Population: A total of 1527 infants were randomized to either placebo or extended NVP. 5 of these infants were later found to be infected at the time of randomization (2 in NVP and 3 in Placebo). Thus, only 1522 infants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Nevirapine | Placebo
Number analyzed (Participants) | 759 | 763
participants
  # of infants with HIV infection at 18 months | 16 | 23
  # of infants @ risk for HIV infection at 18 months | 664 | 663
Statistical Analysis 1: Comparison: Nevirapine; The cumulative rate of HIV infection at 18 months in the extended NVP arm was calculated using the Kaplan-Meier method; while the 95% confidence interval was calculated using Greenwood's formula; Test type: Superiority or Other; Kaplan-Meier Method; 18 mon. Rate of Cum HIV Infection (%) = 2.2, 95% CI 2-sided [1.1 to 3.3]
Statistical Analysis 2: Comparison: Placebo; The cumulative rate of HIV infection at 18 months in the placebo arm was calculated using the Kaplan-Meier method; while the 95% confidence interval was calculated using Greenwood's formula; Test type: Superiority or Other; Kaplan-Meier Method; 18 mon. Rate of Cum. HIV Infection (%) = 3.1, 95% CI 2-sided [1.9 to 4.4]
Statistical Analysis 3: Comparison: Nevirapine vs Placebo; The cumulative rates of HIV infection at 18 months were calculated using the Kaplan-Meier method and were compared between arms using a Z statistic; Test type: Superiority or Other; p = 0.280, Z-test — P-value was not adjusted for interim analysis or multiple testing; Z statistic = 1.081

5. Secondary Outcome: Infant Survival Rates (Mortality Regardless of HIV Infection) in the Two Arms
Time Frame: At Month 18
Measure: Number; unit: participants
Arm/Group | Nevirapine | Placebo
Number analyzed (Participants) | 759 | 763
participants
  # Infant Deaths at 18 months | 26 | 30
  # Infants at risk of death at 18 months | 678 | 684
Statistical Analysis 1: Comparison: Nevirapine; Test type: Superiority or Other; Kaplan-Meier Method; Cumulative Mortality Rate at 18mon (%) = 4.7, 95% CI 2-sided [2.0 to 7.4]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; Kaplan-Meier Method; Cumulative Mortality Rate at 18mon (%) = 4.1, 95% CI 2-sided [2.7 to 5.6]
Statistical Analysis 3: Comparison: Nevirapine vs Placebo; The cumulative rates of mortality at 6 months, as calculated by Kaplan-Meier, were compared between the two groups using a Z-statistic; Test type: Superiority or Other; p = 0.805, Z-test — P-value was not adjusted for interim analysis or multiple testing; Z statistic = -0.247
Statistical Analysis 4: Comparison: Nevirapine; Test type: Superiority or Other; Kaplan-Meier Method; Cumulative Mortality Rate at 6mon (%) = 1.2, 95% CI 2-sided [0.4 to 2.0]
Statistical Analysis 5: Comparison: Placebo; Test type: Superiority or Other; Kaplan-Meier Method; Cumulative Mortality Rate at 6mon (%) = 1.1, 95% CI 2-sided [0.3 to 1.8]
Statistical Analysis 6: Comparison: Nevirapine vs Placebo; The cumulative mortality rates at 18 months, as calculated by Kaplan-Meier, were compared between the two groups using a Z statistic; Test type: Superiority or Other; p = 0.719, Z-test — P-value was not adjusted for interim analysis or multiple testing; Z statistic = -0.360
Statistical Analysis 7: Comparison: Nevirapine vs Placebo; We compared the cumulative mortality rates, as calculated using Kaplan-Meier, between the two study groups over all 18 months of the study follow-up using a log-rank test; Test type: Superiority or Other; p = 0.611, Log Rank

ADVERSE EVENTS:
Time Frame: Regardless of seriousness, severity or relatedness all AEs occurring in infants after enrollment (birth) and throughout the duration of the study (18 months) must be recorded.
Description: Non-serious adverse events occurring in an infant between randomization and 8 months of life will be collected on a case report form. Further, Serious AEs and AEs that meet the DAIDS expedited reporting criteria will be reported through case report forms throughout the entire 18 month follow-up period.
Arm/Group | Nevirapine | Placebo
Serious Adverse Events (participants affected / at risk) | 152/758 | 141/761
Other Adverse Events (participants affected / at risk) | 614/758 | 618/761
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nevirapine (N=758) | Placebo (N=761)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess bacterial (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aneamia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 2 (2) | 4 (7)
Bronchopneumonia (Infections and infestations) | 18 (19) | 20 (23)
Cardipulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cerebral malaria (Infections and infestations) | 1 (2) | 0 (0)
Cerebral palsy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Congenital absence of bile ducts (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Death (General disorders) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 5 (5)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Febrile convulsion (Nervous system disorders) | 5 (5) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 45 (50) | 50 (58)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site abscess (Infections and infestations) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Kwashiorkor (Metabolism and nutrition disorders) | 5 (5) | 9 (9)
Lobar pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 6 (6) | 1 (2)
Malaria (Infections and infestations) | 42 (50) | 34 (40)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Marasmus (Metabolism and nutrition disorders) | 3 (3) | 4 (5)
Measles (Infections and infestations) | 3 (3) | 3 (3)
Meningitis (Infections and infestations) | 2 (2) | 3 (3)
Meningitis bacterial (Infections and infestations) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
Oedema (General disorders) | 1 (1) | 0 (0)
Pericarditis tuberculous (Infections and infestations) | 1 (1) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 20 (21) | 29 (29)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 9 (12)
Sepsis neonatal (Infections and infestations) | 0 (0) | 1 (1)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 3 (4) | 2 (2)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Sudden infant death syndrome (General disorders) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Tonsilitis (Infections and infestations) | 0 (0) | 1 (1)
Traumatic shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nevirapine (N=758) | Placebo (N=761)
Anaemia (Blood and lymphatic system disorders) | 42 (48) | 51 (55)
Conjunctivitis (Eye disorders) | 62 (66) | 43 (53)
Conjunctivitis bacterial (Infections and infestations) | 76 (86) | 72 (80)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 55 (60) | 37 (44)
Diarrhoea (Gastrointestinal disorders) | 57 (63) | 55 (65)
Gastroenteritis (Infections and infestations) | 188 (268) | 208 (288)
Haemoglobin decreased (Investigations) | 73 (76) | 64 (67)
Malaria (Infections and infestations) | 122 (164) | 112 (160)
Neutrophil count decreased (Investigations) | 145 (181) | 121 (153)
Oral candidiasis (Infections and infestations) | 97 (121) | 79 (93)
Upper respiratory infection (Infections and infestations) | 135 (159) | 187 (223)

LIMITATIONS AND CAVEATS:
The rate of maternal highly active antiretroviral therapy use was higher than expected in our study. Thus there were fewer infant infections which decreased the power to detect differences in HIV transmission risks between study groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) & company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review & comment. The publication or other disclosure can be delayed for up to thirty additional business days for manuscripts & five business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.